CLINICAL TRIAL: NCT06698367
Title: Addition of Unilateral Training of the Uninjured Limb to Standard Rehabilitation on Grip Strength and Manual Dexterity of Patients with Surgically Treated Distal Radius Fracture.
Brief Title: Unilateral Training of the Uninjured Limb on Clinical Outcomes in Patients with Surgically Treated Radius Fracture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Catolica de Temuco (Other)
Responsible Party: Principal Investigator, Iván Alejandro Cuyul Vásquez, Principal Investigator, Universidad Catolica de Temuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT-EdCruzada2024
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Wrist Fractures; Distal Radius Fractures
Keywords: Distal radius fracture; Cross-education; Rehabilitation; Exercise
MeSH Terms: conditions — Wrist Fractures; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Opaque sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard rehabilitation plus unilateral high-intensity strength exercise (Experimental): Participants will undergo progressive strength training based on eccentric contractions during the mobilization and strengthening phases of standard rehabilitation.
  Interventions: Other: Standard rehabilitation; Other: Unilateral high-intensity strength exercise
- Standard rehabilitation plus unilateral mobility exercises (Active Comparator): Participants will undergo active mobility training of the pronation-supination movements during the mobilization and strengthening phases of standard rehabilitation
  Interventions: Other: Standard rehabilitation; Other: Unilateral mobility exercises

INTERVENTIONS:
Other: Standard rehabilitation — Protocol based on the best available evidence and to be used in all participants in both groups. The standard rehabilitation protocol will consist of three postoperative phases: Mobilization (0 to 4 weeks), Strengthening (4 to 8 weeks) and Functional phase (8 to 12 weeks). Sessions will be held 3 times a week for 12 weeks. Each session will last 1 hour and will consist of different modalities of therapeutic exercise and cryotherapy.
Other: Unilateral high-intensity strength exercise — Participants will be seated in an armchair with armrests and will perform 4 sets of 8 repetitions of an eccentric exercise for the pronosupinator muscles with a dumbbell with adjustable weights. The training will start with an intensity of 60% of 1RM, until reaching 80% 1RM.
  Arms: Standard rehabilitation plus unilateral high-intensity strength exercise
Other: Unilateral mobility exercises — Participants will be seated in an armchair with armrests and will perform 4 sets of 8 repetitions of an active mobility exercise for the pronation-supination muscles using a plastic rod.
  Arms: Standard rehabilitation plus unilateral mobility exercises

SUMMARY:
The objective will be to determine the effectiveness of adding unilateral upper limb postoperative training to standard rehabilitation compared to standard rehabilitation on maximum grip strength and manual dexterity in patients aged 30-50 years with surgically treated distal radius fracture. It is presumed that the addition of unilateral upper limb training will significantly improve maximum grip strength and manual dexterity at the end of the intervention period compared to the group receiving only standard rehabilitation.

Patients who agree to participate in this research will be randomly assigned to a control group (standard rehabilitation with unilateral training with mobility exercises) or an experimental group (standard rehabilitation with unilateral high-intensity strength training). The duration of the postoperative intervention will be 12 weeks. The primary variables are maximum grip strength and manual dexterity. Secondary variables are wrist mobility, forearm circumference, maximum voluntary isometric strength, functionality and health-related quality of life. Results will be measured at 0, 6 and 12 weeks postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30-50 years
* Radiological diagnosis of unilateral distal radius fracture without concomitant fractures.
* Fracture treated surgically.

Exclusion Criteria:

* Patients with lesion of the triangular fibrocartilage.
* Patients with distal radius fracture with consolidation disorders.
* Patients with health conditions that cause pain or affect the motor skills of the upper limb (radiocarpal osteoarthritis, carpal tunnel syndrome, Quervain's tenosynovitis, neurodegenerative diseases, sequelae of stroke)
* Patients with multi-site pain or chronic polyarticular diseases such as osteoarthritis or rheumatoid arthritis.
* Unstable cardiovascular, respiratory, systemic or metabolic conditions that do not allow high-intensity physical exercise.
* Patients who are taking nutritional supplements that interfere with the regulation of skeletal muscle strength and mass (example: whey protein, creatine, etc.)
* Inability to understand, read and/or speak the Spanish language.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength | 0, 6 and 12 weeks
  Jamar grip dynamometer (kilos)
Manual dexterity | 0, 6 and 12 weeks
  Functional Dexterity Test (Seconds)

SECONDARY OUTCOMES:
Active range motion | 0, 6 and 12 weeks
  Wrist and forearm: Extension, flexion, pronation and supination (degree)
Pain intensity | 0, 6 and 12 weeks
  Visual Analogue Scale (0-10 centimeters)
Forearm circumference | 0, 6 and 12 weeks
  Circumference (cm)
Maximum voluntary isometric strength. | 0, 6 and 12 weeks
  Progressor 300, Tindeq, Norway (Kilos)
Self-reported upper limb function. | 0, 6 and 12 weeks
  Quick Disabilities of Arm, Shoulder and Hand (0-100 points)
Self-reported wrist function | 0, 6 and 12 weeks
  Patient-Rated Wrist Evaluation (0-50 points)
Health-related quality of life | 0, 6 and 12
  Short Form-12 (0-100 points)

OTHER OUTCOMES:
Depression, anxiety and stress | 0 week
  Depression, Anxiety and Stress Scale (0-63 points)
Treatment expectations | 0 week
  Treatment Expectation Questionnaire (0-10 points)
Physical activity | 0 and 12 weeks
  International Physical Activity Questionnaire (Categorical Score: Low, Moderate. High)

CONTACTS AND LOCATIONS:
Locations (1):
- Red Salud, Temuco, Temuco, Chile

IPD SHARING:
Plan to Share IPD: No